CLINICAL TRIAL: NCT01997905
Title: Feasibility Clinical Investigation of a Minimally Invasive Surgically Deployed AtriCure AtriClip Left Atrial Appendage Exclusion System for Stroke Prophylaxis in Patients With Non-Valvular Atrial Fibrillation and in Whom Long Term Oral Anticoagulation Therapy is Medically Contraindicated
Brief Title: Stroke Feasibility Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2011-2
Record Dates: First submitted 2013-11-21; First posted 2013-11-28 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Atrial Fibrillation; AFib
Keywords: Left Atrial Appendage; LAA; Atrial Fibrillation; AFib; AF; IRB approved; clinical; Stroke; TIA; contraindication to oral anticoagulation therapy; Arrhythmias, Cardiac; OAC; trial; study; LAA occlusion; occluded; prevent
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Arrhythmias, Cardiac; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AtriClip LAA Exclusion Device (Experimental): AtriClip delivered via minimally invasive surgical procedure
  Interventions: Device: AtriClip LAA Exclusion Device

INTERVENTIONS:
Device: AtriClip LAA Exclusion Device
  Other Names: LAAØ; PRO1; AtriClip™ LAA Exclusion System; AtriClip™ LAA Exclusion System w/ preloaded Gillinov-Cosgrove™ Clip; AtriClip LAA Exclusion System and Delivery System (LAAØ); AtriClip LAA Exclusion System and Delivery System (PRO1)

SUMMARY:
This is a feasibility study to assess the safety and efficacy of the AtriCure AtriClip when placed via Minimally Invasive Surgical Deployment to the Left Atrial Appendage. The purpose is for evaluation of Stroke Prevention in Patients with Non-Valvular Atrial Fibrillation who are unable to take Oral Anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years and ≤ 80 years of age.
2. Patient has electrocardiographically confirmed non-valvular atrial fibrillation (paroxysmal, persistent, or longstanding persistent AF).
3. CHADS2 or CHA2DS2VASc score ≥2.
4. Patient has medical contraindication to long term anticoagulant therapy (OAC), defined as one or more of the following:

   * history of intracranial bleeding (e.g. due to amyloid angiopathy or other condition) which renders patient unsafe for OAC;
   * history of gastrointestinal, genitourinary, or respiratory tract bleeding due to permanent condition which renders patient unsafe for OAC;
   * HAS-BLED Score ≥ 3.
5. Patient is considered an acceptable surgical candidate, including use of general anesthesia.
6. Female patients must be of non-child bearing potential, or have a negative pregnancy test within 7 days prior to index procedure.

Exclusion Criteria:

1. Stroke within 30 days, or TIA within 3 days, respectively, prior to index procedure.
2. Documented medical history of any penetrating trauma to thorax, or blunt trauma to thorax which resulted in a left pneumothorax or left hemothorax.
3. Myocardial infarction within 60 days prior to index procedure.
4. NYHA Class IV heart failure.
5. Ejection fraction < 40% (based on baseline transthoracic echocardiography (TTE)).
6. Prior attempted obliteration of left atrial appendage (percutaneous or open cardiac surgery).
7. Previous catheter ablation with perforation or complication.
8. Prior open cardiac surgery, or percutaneous coronary intervention with associated unintended cardiac perforation, or pericardial adhesions are suspected.
9. History of pericarditis or pericardiocentesis.
10. Active infection, septicemia, or fever of unknown origin.
11. Concomitant elective surgical procedure (in addition to AtriClip placement) at the time of index procedure.
12. Planned atrial arrhythmia ablation procedure within six months following index procedure.
13. Underlying structural heart disease requiring planned surgical treatment within six months following the index procedure.
14. Cardiac or thoracic surgical procedure within the thirty days prior to index procedure.
15. Anticoagulation therapy for other medical condition (i.e. deep vein thrombosis) is required.
16. Patient unable to discontinue thienopyridines (e.g. clopidogrel) or non-ASA antiplatelet agents 4 days pre-operatively and abstain for at least 2 days post-operatively.
17. Renal Failure as defined by creatinine > 2.0 mg/dl (> 152.5 umol/L) and/or need for dialysis.
18. Known carotid artery diameter stenosis greater than 80%.
19. Patient has symptomatic or high-grade carotid disease (>70% bilaterally).
20. Patient unable or unwilling to undergo transesophageal echocardiography (TEE).
21. Presence of thrombus in the left atrium or LAA, as determined by baseline TTE or Computed Tomography Angiogram (CTA).
22. Documented history of thrombophilic disorder, with diagnosis established via previous objective testing (e.g. familial screening for thrombophilia).
23. Moderate to Severe Chronic Obstructive Pulmonary Disease (FEV1 or VC<70% predicted) or intolerant of single lung ventilation.
24. History of Hypercoagulopathy
25. Body Mass Index (BMI) > 35.
26. Other medical illness or comorbidity that may cause non-compliance with the protocol, confound data interpretation (e.g. severe dementia), or limited life expectancy (i.e. < 3 months).
27. Enrolled in another investigational device or drug study at the time of enrollment and during the course of the study.
28. Psychiatric disorder which in the judgment of the investigator could interfere with informed consent, completion of tests, therapy, or follow-up.
29. Patient is pregnant or intends to become pregnant within 6 months post-index procedure.

Intraoperative Exclusion Criteria

1. Left atrial appendage width < 29mm or > 50mm, based on TEE imaging.
2. Presence of thrombus in the left atrium or LAA based on TEE imaging.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Basel Ramlawi, MD, Principal Investigator — Methodist Hospital Houston
Locations (7):
- United States (7):
  - St. Helena Hospital, St. Helena, California
  - Mercy Hospital, Miami, Florida
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Houston Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Aspirus, Wausau, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled (defined as signed informed consent) on March 25, 2014. The last subject completed their final visit as of July 31, 2015. A total of 13 subjects were enrolled from 4 sites. Of the 13 enrolled subjects, 10 were treated (defined as attempted surgery) with the investigational device.
Groups:
- AtriClip LAA Exclusion Device: AtriClip delivered via minimally invasive surgical procedure
  AtriClip LAA Exclusion Device
Period: Overall Study
Arm/Group | AtriClip LAA Exclusion Device
Started | 13
Baseline Completed | 11
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72 (8.85)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
NYHA Functional Class [Number; unit: participants] — Doctors usually classify patients' heart failure according to the severity of their symptoms. The table below describes the most commonly used classification system, the New York Heart Association (NYHA) Functional Classification. It places patients in one of four categories based on how much they are limited during physical activity(http://www.heart.org/HEARTORG/Conditions/HeartFailure/AboutHeartFailure/Classes-of-Heart-Failure_UCM_306328_Article.jsp#.V8WM3md4epo). The higher the category, the more severe the symptoms.
  participants
    I (No symptoms and no limitations) | 6
    II (Mild symptoms and slight limitation) | 3
    III (Marked limitation) | 0
    IV (Severe limitations) | 0
    No Heart Block | 1
    Not Reported | 1
CHADS2 Score [Mean (Standard Deviation); unit: units on a scale] — CHADS2 is based on the following: Congestive Heart Failure, Hypertension, Age (75 years or older), Diabetes Mellitus, and Stroke (history of stroke or transient ischemic attack). For each factor that is present, the patient receives one point for a total of 6 points. The higher the CHADS2 score the higher the stroke risk.
  units on a scale | 2.9 (0.88)
CHA2DSVAS Score [Mean (Standard Deviation); unit: units on a scale] — CHA2DS2-VASc included additional 'stroke risk modifier' risk factors to the CHADS2. CHA2DS2-VASc score was extended to include: age 65-74, female gender and vascular disease. In the CHA2DS2-VASc score, 'age 75 and above' also has extra weight, with 2 points. The maximum CHA2DS2-VASc score is 9 (for age, either the patient is ≥75 years and gets two points, is between 65-74 and gets one point, or is under 65 and get no point). The higher the CHA2DS2-VASc score, the higher the stroke risk.
  units on a scale | 4.6 (0.84)
HAS-BLED Score [Mean (Standard Deviation); unit: units on a scale] — A risk score to estimate the one year risk of major bleeding (i.e. intracranial, requiring hospitalization, hemoglobin decrease> 2g/L, and/or transfusion) in patients with atrial fibrillation. HAS-BLED score can range from 0 to 9 points, depending upon the number of risk factors for a given patient. HAS-BLED includes the following factors: Hypertension, Abnormal Kidney and/or Liver Function, Stroke (previous history of stroke, especially deep brain (lacunar) stroke), Bleeding, Labile INR, Elderly (>65 years) and Drugs and/or alcohol. The higher the score, the higher the risk of bleeding.
  units on a scale | 3.6 (0.70)

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events Within 30 Days Post-Index Procedure
Description: The primary safety endpoint consists of the following serious adverse events within 30 days post-index procedure (unless otherwise noted), as adjudicated by Independent Physician Adjudicator:
  * Serious Injury to the cardiac structure or other body structure deemed to be related to the delivery or placement of the Clip
  * Cardiac-Related Death, Myocardial Infarction, or Ischemic Stroke
  * Major bleeding (defined as requiring re-operation and/or transfusion (> 2 U packed red blood cells (PRBC)) within any 24 hour period during the first 2 days post-index procedure or at any time point if attributed to the device/index procedure).
Time Frame: 30 days post-index procedure
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 10
participants | 0

2. Primary Outcome: Composite Left Atrial Appendage Placement and Exclusion Success
Description: Primary Efficacy endpoint is a success/failure endpoint with success requiring all of the following:
  1. Patient Technical Success: The ability to successfully implant an AtriClip device at the LAA in a patient.
  2. Intra-Procedural Complete Exclusion of the LAA: The complete exclusion of the LAA defined by lack of fluid communication (<3 mm residual communication with LAA and <10 mm residual pocket) between the LA and LAA, assessed intra-procedurally by TEE.
  3. 3 Month Follow-Up Complete Exclusion of the LAA: The complete exclusion of the LAA defined by lack of fluid communication (<3 mm residual communication with LAA and < 10mm residual pocket) between the LA and LAA at >=3 month TEE or CTA evaluation.
Time Frame: Immediate to 3-months post-index procedure
Population: Ten (10) patients were treated, however the AtriClip® device was not implanted in one (1) patient.
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 9
participants | 8

3. Secondary Outcome: Rate of Stroke and Non-CNS Systemic Embolism
Description: The secondary efficacy endpoints will be a composite of the following events within 3 months and 6 months post-index procedure:
  1. Stroke (ischemic )
  2. Non-CNS (Central Nervous System) systemic embolism.
Time Frame: 3 months and 6 months post-index procedure
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 10
participants | 0

4. Secondary Outcome: Serious Device or Procedure Related Adverse Event Rate
Description: Overall Serious Device or Procedure Related Adverse Event Rate: Incidence of all serious device or procedure related adverse events observed through the 3 month and 6 month follow-up assessments as adjudicated by Independent Physician Adjudicator.
Time Frame: 3 month and 6 month post-index procedure
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 10
participants | 0

5. Secondary Outcome: Overall Serious Adverse Event Rate
Description: Overall Serious Adverse Event Rate: Incidence of all serious adverse events, regardless of attribution, observed through the 3 month and 6 month follow-up assessments, as adjudicated by Independent Physician Adjudicator.
Time Frame: 3 month and 6 month Post Index Procedure
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 10
participants
  Cardiac Disorder | 3
  General Disorder | 1
  Infections and Infestations | 2
  Neoplasms Benign (Carcinoid Tumor Pulmonary) | 1
  Respiratory Failure | 1

6. Secondary Outcome: Overall Adverse Event Rate
Description: Overall Adverse Event Rate: Incidence of all device and procedure related adverse events and any neurological related AEs, regardless of attribution, observed through the 3 month and 6 month follow-up assessments, as adjudicated by Independent Physician Adjudicator.
Time Frame: 3 month and 6 month post-index procedure
Population: All treated patients.
Measure: Number; unit: participants
Arm/Group | AtriClip LAA Exclusion Device
Number analyzed (Participants) | 10
participants
  Blood and Lymphatic System Disorders (Anaemia) | 3
  Cardiac Disorder | 3
  Eye Disorder (Cataract) | 1
  Gastrointestinal Disorder | 3
  General Disorder | 3
  Immune Disorder (Seasonal Allergy) | 1
  Infections and Infestations | 5
  Injury (Accident at Home, Radius Fracture) | 2
  Investigations | 2
  Metabolism and Nutrition Disorder | 1
  Neoplasms Benign (Carcinoid Tumor Pulmonary) | 1
  Nervous System Disorder | 1
  Psychiatric Disorder | 1
  Renal and Urinary Disorder | 2
  Respiratory Disorder | 4
  Surgical and Medical Procedure | 1
  Vascular Disorder | 2

ADVERSE EVENTS:
Time Frame: Incidence of Serious Adverse Events reported during the study
Arm/Group | AtriClip LAA Exclusion Device
Serious Adverse Events (participants affected / at risk) | 5/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriClip LAA Exclusion Device (N=10)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Pnemonia (Infections and infestations) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Carinoid tumor pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriClip LAA Exclusion Device (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Cardiovascular Deconditioning (Cardiac disorders) | 3 (3)
Diastolic Dysfunction (Cardiac disorders) | 1 (1)
Sick Sinus Sundrome (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Chest Pain (General disorders) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Accident at Home (Injury, poisoning and procedural complications) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1)
Biopsy Lung Abnormal (Investigations) | 1 (1)
Troponin Increased (Investigations) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1)
Carinoid Tumor Pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered State of Consciousness (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiatory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No